CLINICAL TRIAL: NCT01457768
Title: A Long Term Follow-up Registry Study of Subjects Who Did Not Achieve Sustained Virologic Response in Gilead-Sponsored Trials in Subjects With Chronic Hepatitis C Infection
Brief Title: A Gilead Sequence Registry of Subjects Who Did Not Achieve Sustained Virologic Response
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-248-0123; 2011-000946-39 (EudraCT Number)
Record Dates: First submitted 2011-10-04; First posted 2011-10-24 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Tegobuvir; Registry; HCV RNA; Treatment experienced; Treatment naive; GS 9451; GS 5885; Sequence; GS 5816; GS 7977; Sofosbuvir; Sovaldi™; SOF; Ledipasvir; LDV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This Registry is designed to obtain long term data on participants who have failed to achieve sustained virologic response (SVR) while receiving at least one Gilead oral antiviral agent (OAV) in a previous Gilead-sponsored hepatitis C virus (HCV) study.

ELIGIBILITY:
Key Inclusion Criteria:

* Have previously participated in a Gilead-sponsored hepatitis C study and received at least one Gilead OAV
* Have failed to achieve an SVR in a previous Gilead-sponsored study, as defined in the original treatment protocol
* Provide written, informed consent
* Be willing and able to comply with the visit schedule

Key Exclusion Criteria:

* Individuals planning to start a new course of hepatitis C therapy including any investigational drug or device during the course of the follow-up Registry
* History of clinically significant illness or any other major medical disorder that may interfere with follow-up, assessments or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have failed to achieve sustained virologic response (SVR) while receiving at least one Gilead OAV in a previous Gilead-sponsored HCV study.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with at least one drug resistant mutation (DRM) loss from enrollment to end of study by treatment regimen | Up to 3 years

SECONDARY OUTCOMES:
Proportion of participants with DRM loss by unit category, 1, 2, 3,…n, by treatment regimen | Up to 3 years
Average number of DRM loss by treatment regimen | Up to 3 years
Liver disease progression | Up to 3 years
  Liver disease progression is a composite endpoint measured by laboratory parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, albumin, platelets, prothrombin time (PT) and α-fetoprotein) and observed or reported clinical signs and symptoms.
Proportion of participants who develop hepatocellular carcinoma (HCC) through Week 144 by treatment regimen | Up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (318):
- United States (156):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Advanced Clinical Research Institute, LLC, Anaheim, California
  - Franco Felizarta, MD, Bakersfield, California
  - Southern California Medical Group, Coronado, California
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - UC Davis Medical Center, Davis, California
  - Kaiser Permanente Institute for Health Research, La Jolla, California
  - Scripps Clinic, La Jolla, California
  - University of California San Diego, La Jolla, California
  - eStudySite, La Mesa, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Kaiser Permanente of Colorado, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - 8631 West 3rd Street, Los Angeles, California
  - California Liver Institute, Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Administration Wadsworth Medical Center, Los Angeles, California
  - eStudySite, Oceanside, California
  - Stanford University, Palo Alto, California
  - 660 South Fair Oaks Avenue, Pasadena, California
  - UC Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Research and Education, Inc., San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - University of California, San Francisco School of Medicine, San Francisco, California
  - San Francisco General Hospital, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - San Jose Gastroenterology, San Jose, California
  - Silicon Valley Research Institute, San Jose, California
  - Los Angeles BioMedical Institute at Harbor-UCLA Medical Center, Torrance, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Pointe West Infectious Diseases d/b/a Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Orlando Immunology Center-, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Saint Joseph's Hospital, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Medical College of Wisconsin, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Community Research Initiative of New England, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Partners in Internal Medicine, PC, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - 200 1st st SW, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Digestive Health Specialists, Tupelo, Mississippi
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Impact Clinical Trials, Las Vegas, Nevada
  - ID Care, Inc., Hillsborough, New Jersey
  - Research Center at Affiliates in Gastroenterology, Morristown, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology Associates, Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - Concorde Medical Group PLLC, New York, New York
  - Weill Medical College of Cornell Univeristy, New York, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai Beth Israel, New York, New York
  - Saint Luke's-Roosevelt Hospital Center, New York, New York
  - University of Rochester, Rochester, New York
  - Westchester Medical Center, Yonkers, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Options Health Research LLC, Tulsa, Oklahoma
  - Schleinitz Research and Gastroenterology LLC, Medford, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Health Network, Network Office of Research and Innovation, Allentown, Pennsylvania
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Center of the MidSouth, P.C., Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Gastro One, Germantown, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - The North Texas Research Institute, Arlington, Texas
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Austin Hospital, Austin, Texas
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Nicholaos C. Bellos, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - University of Utah Pediatric Pulmonology, Salt Lake City, Utah
  - PRA Health Sciences, Salt Lake City, Utah
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Liver Institute of Virginia, Bon Secours Health System, Richmond, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Wisconsin Hospital and Clinic, Madison, Wisconsin
- Australia (19):
  - Canberra Specialist Centre, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - 102 Burton Street, Darlinghurst, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Greenslopes Private Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital - Infectious Disease Unit, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - St Vincent's University Hospital, Fitzroy
  - Royal Brisbane & Women's Hospital, QLD
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Wilhelminenspital der Stadt Wien, Vienna, Vienna
- Canada (12):
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - Inspiration Research Limited, Toronto, Ontario
  - University of Calgary, Calgary
  - University of Alberta, Edmonton
  - Hopital Saint-Luc du CHUM, Montreal
  - Toronto General Hospital, Toronto
  - Toronto Western Hospital, Toronto
  - LAIR Centre, Vancouver
  - Gordon & Leslie Diamond Health Care Centre, Vancouver
  - University of British Colombia, Vancouver
  - GIRI GI Research Institute, Vancouver
  - University of Manitoba, Health Sciences Center, Winnipeg
- Czechia (2):
  - Klinmed, s.r.o., Prague
  - Remedis, s.r.o., Nestátní zdravotnické zarízení, Vladimírova 10, Prague
- Estonia (2):
  - West Tallinn Central Hospital, Talinn
  - Tartu University Hospital, Tartu
- France (20):
  - Hôpital Haut-Lévêque, CHU Bordeaux, Pessac, Aquitaine
  - Centre Hospitalier Universitaire de Grenoble, Cedex 9, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - Service des Maladies de l'Appareil Digestif et de la nutrition, Lille, Hauts-de-France
  - Hôpital Claude Huriez- Service d'Hépato-Gastroentérologie, Lille, Hauts-de-France
  - Hôpital-Saint Joseph, Service D'Hépato-Gastroentérologie, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital de I´Archet 2, Nice, Provence-Alpes-Côte d'Azur Region
  - Hopital Beaujon, Clichy
  - Hopital Saint-Eloi, Montpellier
  - CHU de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint Louis, Services des Maladies Infectieuses, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Pontchaillou, Rennes
  - C.H.U. Strasbourg - Hôpital Hautpierre - Hématologie, Strasbourg
  - CHU de Nancy, Vandœuvre-lès-Nancy
  - Hôpital Henri Mondor, Créteil, Île-de-France Region
  - Service Maladies Infectieuses, Paris, Île-de-France Region
  - Hôpital La Pitié Salpétrière, Service des Maladies Infectieuses, Paris, Île-de-France Region
  - Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
- Germany (33):
  - Bertoldstrasse 48, Freiburg im Breisgau, Baden-Wurttemberg
  - Albert-Ludwigs-Universität, Freiburg im Breisgau, Baden-Wurttemberg
  - Medizinische Universitätsklinik IV (Krehl Klinik) Abt. Gastroenterologie und Infektionskrankhen, Heidelberg, Baden-Wurttemberg
  - Infektiologikum, Frankfurt am Main, Hesse
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - CRC Hannover, Hanover, Lower Saxony
  - Klinik für Gastroenterologie und Hepatologie am Abdominalzentrum, Cologne, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Medizinisches Zentrum - Klinik für Gastroenterologie und Hepatologie, Essen, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis, Herne, North Rhine-Westphalia
  - Leber- and Studienzentrum am Checkpoint, Berlin
  - Charite Campus Virchow-Klinikum, Berlin
  - Seestrasse 13, Berlin
  - MIB Dienstleistung GmbH, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Klinikum der Johann Wolfgang-Goethe-Universität, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Universitatsklinik, Freiburg im Breisgau
  - Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Institut für interdisziplinäre Medizin Studien GmbH an der Asklepiosklinik Saint Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Universität Heidelberg, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Kiel, Kiel
  - University of Leipzig, Leipzig
  - Johannes Gutenberg University Hospital, Mainz
  - Mainz University, Mainz
  - Klinikum Innenstadt der LMU Munchen, München
  - Universitätsklinik Würzburg, Wüerzburg
  - Universitätsklinikum Würzburg - Med Klinik und Poliklinik, Würzburg
- Italy (16):
  - Casa Sollievo della Sofferenza Hospital, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospedaliera S. Orsola - Malpighi, Bologna
  - Ente Ospedaliero Ospedali Galliera di Genova, Genova
  - Ospedale San Raffaele-IRCCS, Centro San Luigi - San Raffaele Turro, Unità Operativa di Malattie Infettive, Milan
  - Azienda Ospedaliera, Milan
  - Dipartimento Polispecialistico - Malattie Infetive, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Padova, U.O.C. Cardiologia, Padua
  - Azienda Ospedaliera-universitaria Policlinico P. Giaccone, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Malattie Infettive - Epatologia, Roma
  - Fondazione Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Universitair Medisch Centrum Sint Radboud, Nijmegen
- New Zealand (9):
  - Auckland Clinical Studies Limited, Grafton, Auckland
  - Middlemore Hospital, Grafton, Auckland
  - Auckland City Hospital, Grafton, Auckland
  - Bay of Plenty Clinical School, Tauranga, Bay of Plenty
  - Wellington Hospital, Newton, WGN
  - Christchurch Hospital, Christchurch
  - Waikato Hospital (District Health Board), Hamilton
  - Urosurgery, Hamilton
  - Wellington Hospital, Wellington
- Poland (10):
  - Centrum Badan Klinicznych Osrodek Badan Wczesnej Fazy, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - Oddzial Dzienny, Warsaw, Masovian Voivodeship
  - SP ZOZ Wojewódzki Szpital Zakazny, Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Kazimierza Dluskiego w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Szpital Specjalistyczny w Chorzowie, Chorzów, Silesian Voivodeship
  - ID Clinic, Mysłowice, Silesian Voivodeship
  - SP ZOZ Wojewodzki Szpital Zakazny w Warszawie, Chorzów
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Lodz
  - NZOZ Pol-SaNa-Med, Mysłowice
- Puerto Rico (3):
  - Chattanooga Hem/Oncology Ass (SCRI), San Juan, PR
  - Clinical Research Puerto Rico, San Juan, PR
  - Fundacion De Investigacion De Diego, San Juan
- Spain (11):
  - C / Manuel de Falla, Majadahonda, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Moncloa, Servicio de Enfermedades Infecciosas, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Paseo de la Castellana nº 261, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Avenida Tres Cruces s/n, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset, Östra sjukhuset, Gothenburg, Västra Götaland County
  - Sahlgrenska Universitetssjukhuset, Östra Sjukhus, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Skånes Universitetssjukhus i Lund, Lund
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska Universitetssjukhuset Solna, Solna
- United Kingdom (13):
  - University of Birmingham and Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Southampton University Hospitals NHS Trust, Southampton General Hospital, Hampshire, England
  - Westminster Bridge Road, London, England
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - Guy's and Saint Thomas NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - King's College Hospital, London, England
  - St George Hospital, London, England
  - North Manchester General Hospital, Manchester, England
  - Queen's Medical Centre Campus, Nottingham, England
  - John Radcliffe Hospital, Oxford, England
  - Marlborough Street, Bristol
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Younossi ZM, Stepanova M, Racila A, Afendy A, Lawitz EJ, Schwabe C, Ruane PJ, Lalezari J, Reddy KR, Jacobson IM, Muir AJ, Gaggar A, Myers RP, Younossi I, Nader F. Long-term Benefits of Sustained Virologic Response for Patient-Reported Outcomes in Patients With Chronic Hepatitis C Virus Infection. Clin Gastroenterol Hepatol. 2020 Feb;18(2):468-476.e11. doi: 10.1016/j.cgh.2019.07.047. Epub 2019 Jul 31. PMID 31376493
- [Derived] Younossi ZM, Stepanova M, Jacobson I, Muir AJ, Pol S, Zeuzem S, Younes Z, Herring R, Lawitz E, Younossi I, Racila A. Not Achieving Sustained Viral Eradication of Hepatitis C Virus After Treatment Leads to Worsening Patient-reported Outcomes. Clin Infect Dis. 2020 Feb 3;70(4):628-632. doi: 10.1093/cid/ciz243. PMID 30949674